CLINICAL TRIAL: NCT07035067
Title: Multidimensional Burden of Platinum Resistant Ovarian Cancer (PROC) on Patients and Caregivers in Canada
Status: Enrolling by invitation | Type: Observational
Sponsor: PeriPharm (Other)
Responsible Party: Sponsor
Other Study IDs: Ovarian Cancer
Record Dates: First submitted 2025-06-04; First posted 2025-06-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Caregiver Burden; Patient Burden
MeSH Terms: conditions — Ovarian Neoplasms; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with PROC part of Ovarian Cancer Canada mailing lists
  Interventions: Other: No intervention
- Caregiver of PROC patients part of Ovarian Cancer Canada mailing lists
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No specific intervention is assess in this study.

SUMMARY:
Filling the gap in Canadian evidence on the burden of PROC on QoL is essential. It will help better understand the impact of PROC on multiple aspects of the lives of patients and their caregivers and the real-life hurdles faced by PROC patients and their caregivers. The outputs of this study will help better understand the hurdles and challenges they face and the significant unmet medical need.

ELIGIBILITY:
Patient Inclusion Criteria

1. ≥18 years old
2. Patients with PROC who received >1 prior line of therapy identified through a screening survey. PROC will be defined as recurrence less than 6 months after last platinum chemotherapy (i.e. carboplatin or cisplatin)
3. Ability to read and understand French or English
4. Signature of ICF

Patients Exclusion Criteria

1. Patients with PSOC, defined as those who:

   1. Have not progressed within less than 6 months after completion of platinum-based chemotherapy or;
   2. Are still on platinum chemotherapy or;
   3. Receive maintenance therapy.
2. Patients with platinum-refractory ovarian cancer, defined as not responding or disease progressing during therapy or within three months after the last dose

Caregivers Inclusion Criteria:

1. ≥18 years old
2. Current caregiver of a patient with PROC (see definition to be used above) who received >1 prior line of therapy identified through a screening survey.
3. Ability to read and understand French or English
4. Signature of ICF.

Caregivers Exclusion Criteria:

1. Caregivers of patients with PSOC (see definition above)
2. Caregivers of PROC patients who have passed away
3. Caregivers of platinum-refractory patients (see definition above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer and caregivers of patients with ovarian cancer who are part Ovarian Cancer Canada mailing list.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To estimate the quality of life of patient with ovarian cancer | At recruitment
  Using the the Functional Assessment of Cancer Therapy - Ovarian (FACT-O) and EuroQol 5-dimendion 5-level (EQ-5D-5L)

SECONDARY OUTCOMES:
Patient's symptoms assessment | At recruitment
  Using the Measure of Ovarian Symptoms and Treatment (MOST-T24 (V2))
Caregiver's Quality of Life | At recruitment
  Using the CareGiver Oncology Quality of Life (CarGOQoL) questionnaire
Patients and caregivers work productivity loss and activity impairment | At recruitment
  Using the Work Productivity and Activity Impairment (WPAI) questionnaire
Patient's preference in treatment | At recruitment
  Using a questionnaire specifically developed for this study based on a literature search, physician input and patient association input.

CONTACTS AND LOCATIONS:
Locations (1):
- PROxy Network, an initiative of PeriPharm Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No